CLINICAL TRIAL: NCT02618928
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in France
Brief Title: The Effectiveness of Paritaprevir/Ritonavir - Ombitasvir, ± Dasabuvir, ± Ribavirin in France
Acronym: OPALE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-405
Record Dates: First submitted 2015-11-24; First posted 2015-12-02 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-02

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 8, 12, or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
  The prescription of treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, and was made independently from this observational study and preceded the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
This study seeks to determine the effectiveness of the interferon-free ABBVIE REGIMEN ± ribavirin (RBV) in participants with chronic hepatitis C (CHC) virus in clinical practices across France.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced participants with confirmed CHC, genotype 1 or 4
* Participants receiving or who will receive the interferon-free ABBVIE REGIMEN ± RBV according to product label
* RBV prescribed in line with the current local label

Exclusion Criteria:

* Participant is not participating or intending to participate in a concurrent interventional therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients chronically infected with HCV, receiving the interferon-free ABBVIE REGIMEN, were offered the opportunity to participate in this study during a routine clinical visit at the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 735 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (70):
- France (70):
  - Hopital Saint Joseph /ID# 144927, Marseille, Bouches-du-Rhone
  - Hopital Saint Joseph /ID# 145560, Marseille, Bouches-du-Rhone
  - Hopital Saint Joseph /ID# 145571, Marseille, Bouches-du-Rhone
  - CHR Orleans - Hopital de la Source /ID# 147250, Orléans, Centre-Val de Loire
  - CHU de Besancon - Jean Minjoz /ID# 145884, Besançon, Doubs
  - CHU Dupuytren /ID# 144920, Limoges, Franche-Comte
  - Hopital Universitaire Purpan /ID# 145869, Toulouse, Haute-Garonne
  - Hopital Universitaire Purpan /ID# 150141, Toulouse, Haute-Garonne
  - Hopital Saint Eloi /ID# 144919, Montpellier, Herault
  - Hopital de la Timone /ID# 145558, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital de la Timone /ID# 145574, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU Amiens Picardie /ID# 145871, Amiens, Somme
  - C.H. du Pays d'Aix /ID# 144922, Aix-en-Provence
  - Cabinet medical /ID# 147359, Aix-en-Provence
  - CHU d'Angers /ID# 145880, Angers
  - Centre Hospitalier Victor Dupo /ID# 147241, Argenteuil
  - Centre Hospitalier D'Avignon /ID# 151098, Avignon
  - Centre Hospitalier D'Avignon /ID# 151343, Avignon
  - Cabinet Medical /ID# 147322, Besançon
  - Centre Endo Nord Isere /ID# 148694, Bourgoin
  - Centre Hospitalier Universitai /ID# 147568, Caen
  - CH de Chambery /ID# 145573, Chambéry
  - Hopital Antoine Beclere /ID# 149251, Clamart
  - Hopital Antoine Beclere /ID# 149252, Clamart
  - Centre Hosp Intercommunal /ID# 145876, Créteil
  - Hospital Henri Mondor /ID# 144918, Créteil
  - Clinique du Palais /ID# 145563, Grasse
  - CHU de Grenoble - Albet Michal /ID# 145881, Grenoble
  - CH d'Hyeres /ID# 145870, Hyères
  - Ch Du Mans /Id# 147415, Le Mans
  - Dr. Cuissard, Le Port, FR /ID# 145565, Le Port
  - Centre Hospitalier de Libourne /ID# 145564, Libourne
  - CH Des Deux Vallees Longumeau /ID# 149336, Longjumeau
  - Hopital de la Croix Rousse /ID# 149776, Lyon
  - Ctr Consultations La Sauvegard /ID# 147236, Lyon
  - Hopital de la Timone /ID# 147237, Marseille
  - Ctre Hosp de Montelimar /ID# 147239, Montélimar
  - Cabinet Medical, Boyer Darrigr /ID# 145562, Nanterre
  - CHU de Nice /ID# 144921, Nice
  - Cabinet Medical, Dr. Verdier, /ID# 145575, Nîmes
  - Hopital Saint Antoine /ID# 145567, Paris
  - Hopital Saint Antoine /ID# 148635, Paris
  - Hopital Saint Antoine /ID# 148693, Paris
  - Hopital Saint Antoine /ID# 152825, Paris
  - Cabinet Medical, Giuily /ID# 145882, Paris
  - Hopital Bichat-Claude Bernard /ID# 149246, Paris
  - Cabinet Medical /ID# 145559, Paris
  - Hopital Pitie Salpetriere /ID# 145556, Paris
  - Hopital Pitie Salpetriere /ID# 145566, Paris
  - Hopital Pitie Salpetriere /ID# 149337, Paris
  - Hopital Bichat Claude Bernard /ID# 145886, Paris
  - Hopital Tenon /ID# 145885, Paris
  - CH Marechal Joffre /ID# 145875, Perpignan
  - CHU Jean Bernard /ID# 147414, Poitiers
  - CHU de Reims /ID# 148477, Reims
  - Hospital Pontchaillou /ID# 145883, Rennes
  - Charles Nicolle Hosp chu rouen /ID# 145557, Rouen
  - Institut Arnault Tzanck /ID# 144925, Saint-Laurent-du-Var
  - Hopital Begin /ID# 145872, Saint-Mandé
  - CHU Strasbourg Hautepierre Hos /ID# 147246, Strasbourg
  - Hopital Foch /ID# 147248, Suresnes
  - Cabinet Medical, Dr. Constant, /ID# 145561, Toulon
  - Clinique Amroise Pare /ID# 144924, Toulouse
  - Hopital Joseph Ducuing /ID# 152832, Toulouse
  - Ctre Hospitalier de Tourcoing /ID# 145568, Tourcoing
  - Cabinet Medical, Barbereau /ID# 145874, Tours
  - Hopital Paul Brousse /ID# 145879, Villejuif
  - Hopital Paul Brousse /ID# 147244, Villejuif
  - Hopital Paul Brousse /ID# 147417, Villejuif
  - Hopital Beaujon /ID# 147923, Clichy, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted in 69 medical centers in France experienced in the treatment of chronic hepatitis C (CHC). The first participant entered the study on 15 December 2015, last patient last visit was on 29 March 2018.
Period: Overall Study
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Started | 735
Received Treatment | 728
Completed (HCV ribonucleic acid (RNA) treatment assessment performed at least 10 weeks post-treatment) | 677
Not Completed | 58
Not completed — Failure to Return | 28
Not completed — Insufficient Virological Response | 1
Not completed — Withdrawal by Subject | 2
Not completed — Death | 3
Not completed — Other | 11
Not completed — Missing | 6
Not completed — Treatment Never Started | 7

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 8, 12, or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years | 570
  66 to 84 years | 151
  85 years or older | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 372
  Male | 356
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 577
  Black | 90
  Asian | 28
  Native American | 1
  Other | 32
Years Since Diagnosis of HCV Infection [Mean (Standard Deviation); unit: years] | 13.8 (10.57)
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 78
  Genotype 1a/1b | 3
  Genotype 1b | 427
  Genotype 1d | 1
  Genotype 1e | 2
  Genotype 1l | 1
  Genotype 1, subtype unknown | 1
  Genotype 1/4, subtype unknown | 1
  Genotype 4a | 39
  Genotype 4a/4c/4d | 11
  Genotype 4c | 3
  Genotype 4c/4d | 5
  Genotype 4d | 14
  Genotype 4e | 2
  Genotype 4f | 7
  Genotype 4h | 1
  Genotype 4k | 1
  Genotype 4r | 2
  Genotype 4, subtype unknown | 129
Cirrhosis Status [Count of Participants; unit: Participants]
  No cirrhosis | 520
  Transition to cirrhosis | 97
  Cirrhosis | 111
Pretreatment Status [Count of Participants; unit: Participants]
  Naive | 489
  Experienced | 238
  Missing | 1
HCV RNA Concentration [Median (Full Range); unit: log10 IU/mL] — Population: The core population included all enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
  log10 IU/mL
    number analyzed (Participants) | 720
    (all) | 6.13 [2.32 to 8.24]
Assigned Treatment Regimen [Count of Participants; unit: Participants] — Treatment regimen was assigned by the physician according to local practice and label. Participants could receive two (paritaprevir/ritonavir and ombitasvir) or three (paritaprevir/ritonavir, ombitasvir, and dasabuvir) direct-acting antiviral (DAA) drugs with or without ribavirin (RBV) for 8, 12, or 24 weeks.
  Participants
    2 DAA without RBV for 12 weeks | 4
    2 DAA with RBV for 12 weeks | 209
    3 DAA without RBV for 8 weeks | 95
    3 DAA without RBV for 12 weeks | 334
    3 DAA with RBV for 12 weeks | 84
    3 DAA with RBV for 24 weeks | 2
Co-morbidities [Count of Participants; unit: Participants]
  Any co-morbidity or co-infection | 387
  Human immunodeficiency virus (HIV) co-infection | 13
  Hepatitis B co-infection | 7
  Tuberculosis co-infection | 1
Drug Users [Count of Participants; unit: Participants]
  Psychoactive drug dependency | 45
  Active injection drug use | 5
  Opiate substitution | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug. Participants with missing HCV RNA were counted as virological failure.
Time Frame: 12 weeks after the last dose of study drug (week 20, 24, or 36 depending on the treatment regimen)
Population: The Core population includes enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 720
percentage of participants | 90.7 [88.4 to 92.6]

2. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment
Description: Virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL.
Time Frame: End of treatment (week 8, 12, or 24 depending on the treatment regimen)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 720
percentage of participants | 94.4 [92.5 to 95.9]

3. Secondary Outcome: Percentage of Participants With Sufficient Follow-up Who Achieved Sustained Virological Response 12 Weeks Post-treatment
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
  The Core Population with sufficient follow-up data regarding SVR12 included all core population participants who
  * had evaluable HCV RNA data ≥ 70 days after the last actual dose of the ABBVIE REGIMEN
  * or a HCV RNA value ≥ 50 IU/mL at the last measurement post-baseline
  * or had HCV RNA < 50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥ 70 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to adverse event) or virologic failure.
Time Frame: 12 weeks after the last dose of study drug (week 20, 24, or 36 depending on the treatment regimen)
Population: The Core population with sufficient follow-up data regarding SVR12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 684
percentage of participants | 95.5 [93.6 to 96.8]

4. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as participants with a virologic response (VR; HCV RNA < 50 IU/mL) at end of treatment (EOT) followed by HCV RNA ≥ 50 IU/mL at any time after the end of treatment.
Time Frame: End of treatment (week 8, 12, or 24 depending on the treatment regimen) and up to 24 weeks after the end of treatment.
Population: The Core population with VR at EOT, who completed treatment, and had ≥ 1 HCV RNA measurement ≥ 70 days post-treatment or were a treatment failure between EOT and day 70.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 648
percentage of participants | 1.2 [0.6 to 2.4]

5. Secondary Outcome: Percentage of Participants With Breakthrough
Description: Breakthrough was defined as at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: 8, 12, or 24 weeks (depending on the treatment regimen)
Population: The Core population with virological response on-treatment and with at least one on-treatment measurement thereafter (including EOT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 404
percentage of participants | 0.5 [0.1 to 1.8]

6. Secondary Outcome: Percentage of Participants With Rapid Virological Response at Week 4 (RVR4)
Description: RVR 4 was defined as participants with HCV RNA < 50 IU/mL at week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 720
percentage of participants | 49.0 [45.4 to 52.7]

7. Secondary Outcome: Percentage of Participants With Sufficient Follow-up Who Achieved Sustained Virological Response 24 Weeks Post-treatment (SVR24)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 24 weeks after the last dose of study drug.
  The Core population with sufficient follow-up data regarding SVR24 included all core population participants who
  * had evaluable HCV RNA data ≥ 126 days after the last actual dose of the ABBVIE REGIMEN
  * or a HCV RNA value ≥ 50 IU/mL at the last measurement post-baseline
  * or had HCV RNA < 50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥ 126 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to adverse event) or virologic failure.
Time Frame: 24 weeks after the last dose of study drug (week 32, 36, or 48 depending on the treatment regimen)
Population: The Core population with sufficient follow-up data regarding SVR24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 616
percentage of participants | 94.8 [92.8 to 96.3]

8. Secondary Outcome: Number of Participants in Each Non-response Category 12 Weeks Post-treatment
Description: SVR12 non-response was categorized according to the following:
  * On-treatment virologic failure (breakthrough [at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment] or failure to suppress [each measured on-treatment HCV RNA value ≥ 50 IU/mL]);
  * Relapse, defined as HCV RNA < 50 IU/mL at EOT followed by HCV RNA ≥ 50 IU/mL post-treatment in patients who completed treatment (not more than 7 days shortened);
  * Death
  * Premature treatment discontinuation with no on-treatment virologic failure;
  * Insufficient virological response reported or HCV RNA ≥ 50 IU/mL post-EOT and none of the above criteria
  * Missing SVR12 data and/or none of the above criteria.
Time Frame: 12 weeks after the last dose of study drug (week 20, 24, or 36 depending on the treatment regimen)
Population: The Core population
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 720
Participants
  On-treatment virological failure | 11
  Relapse | 7
  Death | 2
  Premature treatment discontinuation | 14
  Insufficient virological response reported | 3
  Missing/none of the above | 30

9. Secondary Outcome: Percentage of Participants With Adherence to the ABBVIE Regimen, by Adherence Category
Description: Adherence to the ABBVIE treatment regimen is expressed as a percentage of the target dose and was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration) * 100 The ABBVIE regimen consists of paritaprevir/r and ombitasvir with or without dasabuvir.
Time Frame: From first dose of study drug to end of treatment, 8 to 24 weeks depending on the treatment regimen.
Population: Core population
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 720
Participants
  > 105% | 38
  > 95% to ≤ 105% | 623
  > 80% to ≤ 95% | 19
  > 50% to ≤ 80% | 15
  ≤ 50% | 15
  Missing | 10

10. Secondary Outcome: Percentage of Participants With Adherence to Ribavirin by Adherence Category
Description: Adherence to ribavirin is expressed as a percentage of the target dose, and was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration) * 100
Time Frame: From first dose of study drug to end of treatment, 8 to 24 weeks depending on the treatment regimen.
Population: Core population who were prescribed ribavirin
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 292
Participants
  > 105% | 22
  > 95% to ≤ 105% | 219
  > 80% to ≤ 95% | 20
  > 50% to ≤ 80% | 15
  ≤ 50% | 10
  Missing | 6

11. Secondary Outcome: Percentage of Ribavirin Treatment Days in Relation to the Target Number of Ribavirin Treatment Days
Time Frame: From first dose of study drug to end of treatment, 8 to 24 weeks depending on the treatment regimen.
Population: Core population who were prescribed ribavirin and with non-missing data
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 288
percentage of days | 98.5 (13.96)

12. Secondary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medication other than for chronic hepatitis C used from the time when the decision was made to initiate treatment with paritaprevir/ritonavir and ombitasvir with or without dasabuvir until after the last dose.
Time Frame: From first dose of study drug to end of treatment, 8 to 24 weeks depending on the treatment regimen
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 728
Participants
  Any co-medication | 351
  Beta blocking agents | 60
  Analgesics | 58
  Thyroid therapy | 46
  Peptic ulcer / gastro-oesophageal reflux disease | 45
  Benzodiazepine derivatives | 40
  ACE inhibitors | 39
  Diuretics | 37

13. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, or Pregnancies
Time Frame: From first dose of study drug through 30 days after last dose (12 to 28 weeks depending on treatment regimen). The median (minimum, maximum) duration of treatment was 84 (4, 167) days.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 728
Participants
  Any adverse event | 163
  Serious adverse event | 20
  Pregnancy | 1

14. Secondary Outcome: Change From Baseline in Fatigue Impact Scale Total Score
Description: The Fatigue Impact Scale (FIS) questionnaire was used to assess the impact of fatigue on the quality of life of patients.
  The FIS consists of 40 items, each of which is scored 0 (no problem) to 4 (extreme problem), providing a total score from of 0 to 160, where a lower score = less fatigue impact
Time Frame: Baseline, end of treatment (week 8, 12, or 24 depending on the treatment regimen), and at 12 and 24 weeks after end of treatment
Population: Core population with non-missing data at baseline and each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 629
units on a scale
  End of treatment: number analyzed (Participants) | 471
  End of treatment | -6.78 (31.80)
  12 weeks after end of treatment: number analyzed (Participants) | 406
  12 weeks after end of treatment | -18.27 (32.06)
  24 weeks after end of treatment: number analyzed (Participants) | 340
  24 weeks after end of treatment | -16.75 (32.34)

15. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate visual analog scale (VAS).
  Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score by applying country-specific weights.The range for EQ-5D-5L index score is 0 to 1 where '0' is defined as a health state equivalent to being dead and '1' is full health.The higher the score the better the health status.
Time Frame: as for outcome 14
Population: Core population with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 604
units on a scale
  End of treatment: number analyzed (Participants) | 452
  End of treatment | 0.044 (0.208)
  12 weeks after end of treatment: number analyzed (Participants) | 384
  12 weeks after end of treatment | 0.088 (0.202)
  24 weeks after end of treatment: number analyzed (Participants) | 325
  24 weeks after end of treatment | 0.087 (0.196)

16. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) VAS Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status with a separate visual analog scale (VAS).
  The VAS assesses overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: as for outcome 14
Population: Core population with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 630
units on a scale
  End of treatment: number analyzed (Participants) | 476
  End of treatment | 6.8 (18.92)
  12 weeks after end of treatment: number analyzed (Participants) | 407
  12 weeks after end of treatment | 10.6 (17.60)
  24 weeks after end of treatment: number analyzed (Participants) | 350
  24 weeks after end of treatment | 10.4 (17.70)

17. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Absenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Absenteeism indicates the percentage of work time missed due to health problems.
Time Frame: as for outcome 14
Population: The Core population who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 258
percent impairment
  End of treatment: number analyzed (Participants) | 151
  End of treatment | 5.2 (24.2)
  12 weeks after end of treatment: number analyzed (Participants) | 139
  12 weeks after end of treatment | 0.4 (20.5)
  24 weeks after end of treatment: number analyzed (Participants) | 107
  24 weeks after end of treatment | -1.5 (16.8)

18. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Presenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Presenteeism indicates the percentage of impairment while working due to health problems.
Time Frame: as for outcome 14
Population: The Core population who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 259
percent impairment
  End of treatment: number analyzed (Participants) | 148
  End of treatment | -1.2 (28.0)
  12 weeks after end of treatment: number analyzed (Participants) | 137
  12 weeks after end of treatment | -5.5 (25.2)
  24 weeks after end of treatment: number analyzed (Participants) | 105
  24 weeks after end of treatment | -7.4 (22.9)

19. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Work Productivity Impairment (TWP)
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total work productivity impairment (TWP) indicates the percentage of overall work impairment due to health problems.
Time Frame: as for outcome 14
Population: The Core population who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 253
percent impairment
  End of treatment: number analyzed (Participants) | 144
  End of treatment | 1.3 (33.6)
  12 weeks after end of treatment: number analyzed (Participants) | 132
  12 weeks after end of treatment | -4.9 (30.1)
  24 weeks after end of treatment: number analyzed (Participants) | 101
  24 weeks after end of treatment | -8.7 (25.4)

20. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Activity Impairment
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total activity impairment (TAI) indicates the percentage of general (non-work) activity impairment due to health problems.
Time Frame: as for outcome 14
Population: The Core population with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 615
percent impairment
  End of treatment: number analyzed (Participants) | 441
  End of treatment | 1.6 (33.0)
  12 weeks after end of treatment: number analyzed (Participants) | 386
  12 weeks after end of treatment | -7.2 (32.8)
  24 weeks after end of treatment: number analyzed (Participants) | 315
  24 weeks after end of treatment | -9.5 (29.0)

21. Secondary Outcome: Change From Baseline in Beliefs Medication Questionnaire - (18-item BMQ)
Description: The BMQ consists of 2 sections and 18 questions to screen for patients' beliefs, attitudes and concerns about their medication. The BMQ-Specific section comprises two 5-item subscales assessing the necessity of and concerns about the prescribed medication (Specific-Necessity and Specific-Concerns). The BMQ-General section comprises two 4-item subscales assessing beliefs that medicines are harmful and overused by doctors in general (General-Harm and General-Overuse). The 18 items are rated on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). Each subscale score ranges from 1 to 5. High scores in the Specific-Concerns scale represent the notion that adverse reactions are potentially harmful when taking medication on a regular basis, and high scores in the Specific-Necessity scale indicate the patient's need to adhere to medication to maintain health. High scores in the General-Harm and General-Overuse scales represent an overall negative perception of medication.
Time Frame: Baseline and end of treatment (week 8, 12, or 24 depending on the treatment regimen)
Population: The Core population with available data at baseline and end of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 720
units on a scale
  Specific Concerns: number analyzed (Participants) | 445
  Specific Concerns | -0.100 (0.871)
  Specific Necessity: number analyzed (Participants) | 449
  Specific Necessity | -0.099 (0.739)
  General Overuse: number analyzed (Participants) | 477
  General Overuse | 0.119 (0.685)
  General Harm: number analyzed (Participants) | 480
  General Harm | 0.135 (0.670)

22. Secondary Outcome: Change From Baseline in Patient Activation Measure 13 (PAM-13)
Description: PAM 13 is a measure used to assess the patient knowledge, skill, and confidence for self-management, consisting of 13 questions. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4). Scores were summed to calculate the overall raw score, then transformed to a scale with a theoretical range 0 to 100, based on calibration tables, with higher PAM scores indicating higher patient activation.
Time Frame: Baseline and end of treatment (week 8, 12, or 24 depending on the treatment regimen)
Population: The Core population with available data at baseline and end of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 433
units on a scale | 0.44 (9.43)

23. Secondary Outcome: Number of Participants With Outpatient Consultations Due to Liver Disease by Category
Time Frame: as for outcome 13
Population: Core population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 694
Participants
  No outpatient consultations | 515
  One outpatient consultation | 80
  Two or three outpatient consultations | 94
  Four or more outpatient consultations | 5

24. Secondary Outcome: Number of Participants With Hospitalizations Due to Liver Disease by Category
Time Frame: as for outcome 13
Population: Core population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 694
Participants
  No hospitalizations | 685
  One hospitalization | 9

25. Secondary Outcome: Change From Baseline in Percent Glycosylated Hemoglobin (HbA1c)
Time Frame: Baseline and end of treatment (week 8, 12, or 24 depending on the treatment regimen)
Population: Treated participants with available data at baseline and end of treatment.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 17
percent glycosylated hemoglobin | -7.07 (10.70)

ADVERSE EVENTS:
Time Frame: Deaths are reported up to 24 weeks after end of treatment (a maximum of 48 weeks). Adverse events are reported from first dose of study drug through 30 days after last dose (12 to 28 weeks depending on treatment regimen). The median (minimum, maximum) duration of treatment was 84 (4, 167) days.
Groups:
- Paritaprevir/Ritonavir + Ombitasvir Without RBV: Participants received paritaprevir/ritonavir and ombitasvir without ribavirin for either 12 weeks.
- Paritaprevir/Ritonavir + Ombitasvir With RBV: Participants received paritaprevir/ritonavir and ombitasvir with ribavirin for either 12 weeks.
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir without ribavirin for 8 or 12 weeks.
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir with ribavirin for 12 or 24 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir With RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
All-Cause Mortality (participants affected / at risk) | 0/4 | 5/209 | 1/429 | 2/86
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/209 | 13/429 | 6/86
Other Adverse Events (participants affected / at risk) | 1/4 | 33/209 | 38/429 | 11/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir Without RBV (N=4) | Paritaprevir/Ritonavir + Ombitasvir With RBV (N=209) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV (N=429) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV (N=86)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROTHROMBIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAROTID ANEURYSM RUPTURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOMANIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir Without RBV (N=4) | Paritaprevir/Ritonavir + Ombitasvir With RBV (N=209) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV (N=429) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV (N=86)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 22 (22) | 0 (0) | 4 (4)
ASTHENIA (General disorders) | 0 (0) | 6 (6) | 26 (26) | 7 (7)
FATIGUE (General disorders) | 1 (1) | 8 (8) | 12 (12) | 1 (1)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02618928/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT02618928/SAP_001.pdf